CLINICAL TRIAL: NCT06717698
Title: Efficacy, Safety and Pharmacokinetics of NNC0519-0130 Once Weekly s.c. Versussemaglutide 1.0 mg and Placebo in People With Chronic Kidney Disease, With or Without Type 2 Diabetes, and With Overweight or Obesity: a Proof-of-concept and Dose-finding Study
Brief Title: A Research Study Comparing How Well Different Doses of the Medicine NNC0519-0130 Can Reduce Kidney Damage in People Living With Chronic Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9541-7841; U1111-1302-5591 (Other: World Health Organization (WHO)); 2024-510846-15 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Dosing scheme a: NNC0519-0130 (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of NNC0519-0130 following a fixed dose escalation until the maintenance dose is reached.
  Interventions: Drug: NNC0519-0130
- Dosing scheme a: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly.
  Interventions: Drug: Placebo
- Dosing scheme b: NNC0519-0130 (Experimental): Participants will receive once-weekly s.c injections of NNC0519-0130 following a fixed dose escalation until the maintenance dose is reached.
  Interventions: Drug: NNC0519-0130
- Dosing scheme b: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly.
  Interventions: Drug: Placebo
- Dosing scheme c: NNC0519-0130 (Experimental): Participants will receive once-weekly s.c injections of NNC0519-0130 following a fixed dose escalation until the maintenance dose is reached.
  Interventions: Drug: NNC0519-0130
- Dosing scheme c: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly.
  Interventions: Drug: Placebo
- Dosing scheme d: NNC0519-0130 (Experimental): Participants will receive once-weekly s.c injections of NNC0519-0130 following a fixed dose escalation until the maintenance dose is reached.
  Interventions: Drug: NNC0519-0130
- Dosing scheme d: Placebo (Placebo Comparator): Participants will receive NNC0519-0130 matched placebo s.c. once-weekly.
  Interventions: Drug: Placebo
- Dosing scheme e: Semaglutide (Active Comparator): Participants will receive once-weekly s.c injections of semaglutide with a dose escalation done until maintenance dose is reached.
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: NNC0519-0130 — NNC0519-0130 will be administered subcutaneously.
  Arms: Dosing scheme a: NNC0519-0130; Dosing scheme b: NNC0519-0130; Dosing scheme c: NNC0519-0130; Dosing scheme d: NNC0519-0130
Drug: Placebo — Placebo matching NNC0519-0130 will be administered subcutaneously.
  Arms: Dosing scheme a: Placebo; Dosing scheme b: Placebo; Dosing scheme c: Placebo; Dosing scheme d: Placebo
Drug: Semaglutide — Semaglutide will be administered subcutaneously.
  Arms: Dosing scheme e: Semaglutide

SUMMARY:
The study evaluates the safety of different doses of a new medicine called NNC0519 0130. It also looks into how the medicine may improve kidney function in participants with chronic kidney disease with or without type 2 diabetes, living with overweight or obesity. The participants will either get NNC0519-0130 (a new medicine), semaglutide (a medicine that doctors can already prescribe), or placebo (a "dummy" substance). Which treatment the participant will get is decided by chance. The study will last for up to 43 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Female of non-childbearing potential, or male.

  * For US only: Female of childbearing potential using highly effective non-systemic methods of contraception with low user-dependency at least 2 months prior to screening and willingness to continue using it through-out the study, or male.
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus greater than or equal to (≥) 180 days before screening, or not diagnosed with type 2 diabetes mellitus.

  * HbA1c of 6.5 percentage (%)-10.5 percentage (%) [48 - 91 millimoles per mole (mmol/mol)] (both inclusive) if diagnosed with type 2 diabetes mellitus, or HbA1c of less than (<)6.5 percentage (%) [<48 mmol/mol] if not diagnosed with type 2 diabetes mellitus.
* BMI greater than or equal to (≥) 27.0 kilogram per square metre (kg/m^2) at screening.
* Kidney impairment defined by serum creatinine and cystatin C-based Egfr greater than or equal to (≥) 15 and less than (<) 90 mL/min/1.73 m^2.
* Albuminuria defined by Urine Albumin-to-Creatinine Ratio (UACR) greater than or equal (≥)100 and less than (<) 5000 milligram per gram (mg/g).
* Treatment with maximum labelled or tolerated dose of an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB), unless such treatment is contraindicated or not tolerated, in the opinion of the investigator. Treatment dose must be stable for at least 30 days prior to screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective non-systemic contraception with low user-dependency.
* Lupus nephritis or antineutrophil cytoplasmic antibody (ANCA)-associated vasculitis.
* Receiving immunosuppressive therapy for primary or secondary renal disease within 6 months prior to screening.
* Use of any glucagon-like peptide-1 (GLP-1) RA (including medication with GLP-1 RA activity, e.g., GIP/GLP-1 RA) within 90 days prior to screening.
* Myocardial infarction, stroke, transient ischaemic attack, or hospitalization for unstable angina pectoris within 180 days before screening.
* Chronic or intermittent haemodialysis or peritoneal dialysis within 90 days before screening.
* Only applicable for participants with type 2 diabetes (T2D): Uncontrolled and potentially unstable diabetic retinopathy or diabetic maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Presence or history of malignant neoplasms or in situ carcinomas (other than basal or squamous cell skin cancer, low-risk prostate cancer, or in-situ carcinomas of the cervix or carcinoma in situ/high grade prostatic intraepithelial neoplasia (PIN)) within 5 years before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Change in urinary albumin-to-creatinine ratio (UACR) at week 12 | From baseline (week 0) to end of a given maintenance dose period (week 12)
  Measured as a ratio to baseline.
Change in urinary albumin-to-creatinine ratio (UACR) at week 24 | From baseline (week 0) to end of a given maintenance dose period (week 24)
  Measured as a ratio to baseline.
Change in urinary albumin-to-creatinine ratio (UACR) at week 36 | From baseline (week 0) to end of a given maintenance dose period (week 36)
  Measured as a ratio to baseline.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) (creatinine and cystatin C-based Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] 2021) | From baseline (week 0) to end of treatment (week 36)
  Measured in mililitre per minute per 1.73 square metre (mL/min/1.73 m^2).
Change in estimated glomerular filtration rate (eGFR) (creatinine-based CKD-EPI 2021) | From baseline (week 0) to end of treatment (week 36)
  Measured in mililitre per minute per 1.73 square metre (mL/min/1.73 m^2).
Relative change in body weight | From baseline (week 0) to end of treatment (week 36)
  Measured in percentage (%).
Achievement of greater than or equal to (≥) 5 percentage (%) weight reduction | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Achievement of greater than or equal to (≥) 10 percentage (%) weight reduction | From baseline (week 0) to end of treatment (week 36)
  Measured as count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 36)
  Measured in centimetres (cm).
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of a given maintenance dose period (week 12, 24 or 36)
  Measured in percentage point (%-point).
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 36)
  Measured in millimetres of mercury (mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 36)
  Measured in millimetres of mercury (mmHg).
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 40)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (135):
- United States (18):
  - N America Res Inst - San Dimas, San Dimas, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Rocky Mount Reg VA Med-DN, Aurora, Colorado
  - Northeast Research Institute, Fleming Island, Florida
  - Encore Medical Research LLC, Hollywood, Florida
  - Northeast Research Institute, Saint Augustine, Florida
  - Clinical Research of Cent FL, Winter Haven, Florida
  - Endeavor Health, Skokie, Illinois
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - Elite Research Center, Flint, Michigan
  - Clinical Research Consultants, Kansas City, Missouri
  - Albany Medical College, Albany, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Davita Clinical Research, El Paso, Texas
  - Clinical Advancement Center, San Antonio, Texas
  - Tekton Research, San Antonio, Texas
  - Providence Medical Research Center, Spokane, Washington
- Argentina (5):
  - Centro Médico CIMEL, Lanús Este, Buenos Aires
  - Renalida, Mar del Plata, Buenos Aires
  - Centro de Investigaciones Metabólicas, City of Buenos Aires
  - Instituto de Cardiología de Corrientes, Corrientes
  - Instituto de Investigaciones Clinicas Mar Del Plata, Mar del Plata
- Australia (5):
  - Castle Hill Medical Centre, Castle Hill, New South Wales
  - Gosford Renal Research, Gosford, New South Wales
  - Heart of Australia, Chelmer, Queensland
  - Melbourne Renal Research Group, Reservoir, Victoria
  - Sunshine Hospital - Western Centre for Health Research and Education, St Albans, Victoria
- Brazil (6):
  - Quanta Diagnóstico Nuclear / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Instituto Pró-Renal Brasil, Curitiba, Paraná
  - Centro de Diabetes Curitiba, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - Hospital do Rim e Hipertensao Fundacao Oswaldo Ramos, São Paulo
- Bulgaria (8):
  - SRH - Zdrave EAD, Bankya
  - Medical centre Zdrave 1 OOD, Kozloduy
  - Nader Yabrudi - ASMPVBE Individual practice, Smolyan
  - Medical Centre Acad. Iv. Penchev EOOD, Sofia
  - USHATE Akad. Ivan Penchev EAD, Second Clinic of Endocrinology, Sofia
  - UMHAT Sofiamed EAD, Sofia
  - UMHAT Sveta Anna Sofia AD, Second Clinic of Internal Diseases, Sofia
  - UMHAT Sveta Marina EAD, Clinic of Internal Diseases, Varna
- Czechia (8):
  - Nemocnice Český Krumlov, a.s., Český Krumlov
  - MUDr. Petr Buček s.r.o., Frýdek-Místek
  - CTC Hodonin s.r.o., Hodonín
  - FNKV-Internal Clinic-Nephrology, Prague
  - DiaVize s.r.o., Prague
  - IKEM Klinika nefrologie, Prague
  - Fledip s.r.o., Prague
  - Internist Care s.r.o., Smiřice
- India (7):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - MS Ramaiah, Bengaluru, Karnataka
  - Government Medical College, Kozhikode, Kozhikode, Kerala
  - SMS Medical College & Hospital, Jaipur, Rajasthan
  - Diabetes, Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Diabetes Research Center, Hyderabad, Hyderabad, Telangana
  - Nizams Institute of Medical Science, Hyderabad, Telangana
- Italy (8):
  - ASL Avezzano Sulmona L'Aquila - Ospedale San Salvatore - UOC Diabetologia, L’Aquila, Abbruzzo
  - Università degli studi G. D'Annunzio Chieti Pescara - CAST, Chieti, Abruzzo
  - A.O.U. Bologna_ Policlinico S.Orsola Malpighi, Bologna, BO
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Luigi Sacco, Milan
  - Azienda Ospedaliero Universitaria Pisana Ospedale Cisanello, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCS, Roma
- Japan (15):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Fukushima, Japan
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Fujisawa City Hospital_Kidney internal medicine, Kanagawa
  - Higashijujo Sakai Diabetes Clinic_Internal Medicine, Kita-ku, Tokyo
  - Koshigaya Municipal Hospital_Internal medicine, Saitama
  - Hanyu General Hospital_Internal Medicine, Saitama
  - Shinden Higashi Clinic_Internal medicine, Sendai-shi, Miyagi
  - Shinden Higashi Clinic, Sendai-shi, Miyagi
  - Omihachiman Community Medical Center_Nephrology, Siga
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
  - Kato Clinic of Internal Medicine_Internal Medicine, Tokyo
  - Kato Clinic of Internal Medicine, Tokyo
- Malaysia (10):
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Lembah Pantai, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun Ipoh, Ipoh, Perak
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Miri, Miri, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - Hospital Universiti Sains Malaysia, Kota Bharu, Kelantan
  - Prince Court Medical Centre, Kuala Lumpur
  - Hospital Melaka, Malacca
- Poland (17):
  - Kardio Life - Tomasz Borkowski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Terpa Sp. z o.o. Sp. k., Lublin, Lubelskie Voivodeship
  - Kliniczny Szpital Wojewodzki nr 2 im. Sw. Jadwigi Krolowej w Rzeszowie, Rzeszów, Podkarpackie Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Nowy Szpital Sp. z o.o., Gmina Świecie
  - Uniwersyteckie Centrum Kliniczne SUM w Katowicach, Katowice
  - SPZOZ Uniwersytecki Szpital Kliniczny Nr 1 im. Norberta Barlickiego UM w Lodzi, Lodz
  - SP ZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Terpa Sp. z o.o. Sp. k., Lublin
  - Zanamed Medical Clinic Sp. z o.o., Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Formed 2 Sp. z o.o., Oświęcim
  - Uniwersytecki Szpital Kliniczny Nr 2 PUM W Szczecinie, Szczecin
  - Szpitale Tczewskie S.A., Tczew
  - PANSTWOWY INSTYTUT MEDYCZNY MSWiA, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
- South Korea (6):
  - National Health Insurance Corporation Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Pusan National University Hospital, Busan
  - Hallym University Sacred Heart Hospital, Gyeonggi-do
  - Hanyang University GURI Hospital, Gyeonggi-do
  - The Catholic University of Korea, Seoul ST. Mary's Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (8):
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital Universitario de Getafe, Getafe
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Fundacion Jiménez Díaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Clínica Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Universitario Doctor Peset, Valencia
- Turkey (Türkiye) (14):
  - Erciyes Üniversitesi Hastanesi - Nefroloji, Kayseri, Melikgazi
  - Adana Şehir Eğitim ve Araştırma Hastanesi, Adana
  - Hacettepe Universitesi Tip Fakultesi Nefroloji Bilim Dali, Ankara
  - Hacettepe Üniversitesi Hastanesi- Nefroloji, Ankara
  - Ankara Bilkent Şehir Hastanesi-Dahiliye, Ankara
  - Ankara Sehir Hastanesi Dahiliye Klinigi, Ankara
  - Gaziantep Universitesi Tip Fakultesi Hastanesi, Gaziantep
  - Gaziantep Üniversitesi Hastanesi- Endokrinoloji, Gaziantep
  - Göztepe Prof. Dr.Süleyman Yalçın Şehir Hastanesi- Dahiliye, Istanbul
  - T.C SB Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Ege Universitesi Hastanesi- Endokrinoloji, Izmir
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Kocaeli University Nephrology Department, Kocaeli
  - Kocaeli Üniversitesi Araştıma ve Uygulama Hastanesi - Nefroloji, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com